CLINICAL TRIAL: NCT04825561
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel, Phase 3 Clinical Trial to Evaluate the Efficacy and Safety of AD-208 in Male Patients With Androgenetic Alopecia
Brief Title: A Study to Evaluate the Efficacy and Safety of AD-208
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Addpharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AD-208P3
Record Dates: First submitted 2021-03-29; First posted 2021-04-01 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Androgenetic Alopecia
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active Comparator (Active Comparator): AD-208 and Placebo of AD-2081
  Interventions: Drug: AD-208; Drug: placebo of AD-2081
- Placebo Comparator (Placebo Comparator): Placebo of AD-208 and Placebo of AD-2081
  Interventions: Drug: placebo of AD-208; Drug: placebo of AD-2081
- Experimental Comparator (Experimental): Placebo of AD-208 and AD-2081
  Interventions: Drug: AD-2081; Drug: placebo of AD-208

INTERVENTIONS:
Drug: AD-208 — PO, Once daily(QD), 24weeks
  Arms: Active Comparator
Drug: AD-2081 — PO, Once daily(QD), 24weeks
  Arms: Experimental Comparator
Drug: placebo of AD-208 — PO, Once daily(QD), 24weeks
  Arms: Experimental Comparator; Placebo Comparator
Drug: placebo of AD-2081 — PO, Once daily(QD), 24weeks
  Arms: Active Comparator; Placebo Comparator

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of AD-208.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the efficacy and safety of AD-208 in male patients with androgenetic alopecia.

ELIGIBILITY:
Inclusion Criteria:

* Male patients aged 18-50 years, inclusive
* Patients who meet the appropriate criteria according to the classification of hair loss
* Signed informed consent

Exclusion Criteria:

* Patients with hair loss disorders other than androgenetic alopecia
* Other exclusions applied

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 139 (Actual)
Dates: Start 2021-06-09 (Actual); Primary Completion 2023-01-09 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
The amount of Change in the total number of hairs | Baseline, Week 24
  The amount of change in the total number of hairs in the unit area

CONTACTS AND LOCATIONS:
Locations (1):
- The Catholic University of Korea, Eunpyeong St. Mary's Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee S, Kim JE, Lew BL, Huh CH, Kim J, Kwon O, Kim MB, Lee YW, Lee Y, Park J, Kim S, Kim DY, Choi GS, Kang H. Efficacy and Safety of Low-Dose (0.2 mg) Dutasteride for Male Androgenic Alopecia: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Phase III Clinical Trial. Ann Dermatol. 2025 Aug;37(4):183-190. doi: 10.5021/ad.25.048. PMID 40736519